CLINICAL TRIAL: NCT07150325
Title: Integration of Force Control Training and Mirror Visual Feedback on Stroke Patients on Brain Activation and Hand Function
Brief Title: Combination of Force Control Training and Mirror Visual Feedback Device on Stroke Patients on Brain Activation and Hand Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Fong Chin Su, Chair Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A-ER-113-229
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Stroke Patients
Keywords: Hand rehabilitation; Finger force control training; Brain activation; Hand dexterity; Hand strength
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror Visual Feedback Group (Experimental): All the stroke patients were asked to use their unaffected hand to operate the hand training system (TIPr) and place their affected hand behind the mirror on the other hand training system (TIPr). According to the game instructions shown on the tablet screen, they should slowly press the evaluation system with the corresponding fingers of their unaffected hand to reach the target force value. When the unaffected hands started to cooperate with the game instructions, the force exerted by the fingertips will be presented on the tablet, and the mirror would show the mirrored (reflected) image of force output level. The subjects were instructed to keep their eyes contacts on the reflected image from the mirror and simultaneously "imagine" that their affected hand performing the same task as the unaffected hand. Subjects was instructed not to move their affected hand voluntarily.
  Interventions: Device: TIPr; Device: Mirror Visual Feedback Device
- Non-Mirror Visual Feedback Group (Active Comparator): All the subjects were asked to use their unaffected hands to operate the hand training system (TIPr) and place their affected hands behind the mirror on the other hand training system. According to the game instructions shown on the tablet screen, they should slowly press the evaluation system with the corresponding fingers of their unaffected hand to reach the target force value. When the dominant hand starts to cooperate with the game instructions, the force exerted by the fingertips will be presented on the tablet. Different from MVF group, the mirror would be covered. The subjects were instructed to keep their eyes contact on the tablet and imagine the affected hand performing the same task as the unaffected hand without mirror visual feedback. Subjects was instructed not to move their affected hand voluntarily.
  Interventions: Device: TIPr; Device: Mirror Visual Feedback Device(Blocked mirror)

INTERVENTIONS:
Device: TIPr — TIPr is a second-generation device, which is originated from Pressing Evaluation and Training System (PETs), developed by NCKU Motion Analysis Lab. This 2nd generation device is a home-based training device, which equipped with single-axis force sensors and displayed visual feedback through a tablet advantages.
Device: Mirror Visual Feedback Device — A box with two compartments through a partition with two mirrors installed on each side, which is commonly applied in Mirror therapy.
  Arms: Mirror Visual Feedback Group
Device: Mirror Visual Feedback Device(Blocked mirror) — Different from Mirror Visual Feedback Device in MVF group, the mirror was blocked by black curtain or paperboard.
  Arms: Non-Mirror Visual Feedback Group

SUMMARY:
Global elderly population continues to grow. Among the diseases caused by aging, stroke accounts for the highest incidence, and the number of stroke patient is increasing year-by-year. Stroke is a common central nervous system disorder, including infarcts and hemorrhagic strokes. It develops rapidly and causes a wide range of neurological deficits. Clinical manifestations vary depending on the location of the brain damage. Common features include hemiplegia and paresthesia, which may be accompanied by incoordination and speech impairments. This leads to decreased independence in daily life, negatively impacting the quality of life and causing stress for patients and their families.

Hand movements are crucial for 70% of daily activities, yet only approximately 15% of patients can regain normal hand movements. Therefore, hand movement restoration is a key focus of rehabilitation. Previous studies have found that finger pressure training using a hand force control system (Tipr) can improve hand and cognitive function in older adults. However, no studies have examined the effectiveness of this hand force control system in the hemiplegic hand of stroke patients. Mirror therapy, a hand training technique used in stroke rehabilitation, has been shown to improve the function of the hemiplegic limb in stroke patients. However, there are currently no studies examining the application of force control in mirror therapy. Therefore, this study aims to explore and develop a hand rehabilitation method that combines the different compression patterns provided by the hand training system (Tipr) with a mirror training device. By incorporating the mirror's visual feedback of the contralateral limb, the application of the hand training system will be expanded. Non-invasive near-infrared spectroscopy (fNIRs) will be used to assess user brain activation and changes in hand function. This study will investigate user feedback on this rehabilitation method and explore whether force control training can induce bilateral brain interactions and their impact on hand function. The goal is to commercialize this innovative treatment approach for clinical evaluation and training applications.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 20 or older and not participating in any other experimental studies during the study period.
* 2. Patients diagnosed with unilateral cerebral embolism or intracerebral hemorrhage.
* 3. Scores on the Fogel-Meyer Motor Scale-Upper Limb between 20 and 66 (scores indicate poor to full motor function on the affected upper limb), or Brunnstrom stage II or higher for both the proximal and distal upper limbs.
* 4. Mini-Mental State Examination (MMSE) scores, based on educational level: at least 16 for those with no education, at least 21 for those with elementary school education, and at least 24 for those with junior high school education or higher.

Exclusion Criteria:

* 1. Patients with unilateral cerebral hemisphere damage as diagnosed by CT scan.
* 2. Upper limb joint deformity, history of complex or major hand surgery on one hand, or severe hand arthritis.
* 3. Any visual or hearing impairment that would affect experimental performance or prevent compliance with experimental instructions.
* 4. Patients with severe hemispheric neglect.
* 5. Aphasia, which makes it difficult to understand or respond to multiple written or spoken instructions.
* 6. Other factors that may affect participation in the experiment, such as body part loss.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Hand Strength | Before and after intervention(test time:15 minutes)
  Handgrip strength and pinch strength was measured respectively. JAMAR Grip Hand Dynamometer and JAMAR Hydraulic Pinch Gauge were used for the apparatus for force measurement. Pinch strength was divided into lateral pinch, tip pinch and tripod pinch. Each test will test for three times and get the average results.(Adjustable based on stroke patients' hand function) Unaffected hand and unaffected hand need to be evaluated.
Purdue Pegboard Test (PPT) | Before and after intervention(total test time for all subtest: 10 minutes)
  Assess the manual dexterity and coordination for one and both hands, including one hand, two hand and assembly subtest. ( Test for affected hand and unaffected hand). Each subtest test for three times. (Adjustable based on stroke patients' hand function)
Minnesota Manual Dexterity Test (MMDT) | Before and after intervention(total test time for all subtests:25 minutes)
  Assess the eye-hand coordination ability and manual dexterity. MMDT was divided into: Turning, Placing, One hand Turning and Placing, Two hand Turning and Placing, Displacing. (Adjustable based on stroke patients' hand function)
Digit Independence (EN value) | Before and after intervention(test time:40 seconds for each digits)
  The force independence of each digit is collected from the data during force tracking test in evaluation session. The parameter of force independence is an index of five digits overall enslaving presented as EN value. Unaffected hand and unaffected hand need to be evaluated.
Force control ability | Before and after intervention(test time: 40 seconds for each digits)
  Subjects will be asked to track the target force and presses task digit to fit the target line as accurately as possible. Unaffected hand and unaffected hand need to be evaluated.
Oxygenated hemoglobin (HbO) | Before and after intervention(test time:40 minutes or more)
  The Oxygenated hemoglobin (HbO) was measured while the participants play the game under both conditions

SECONDARY OUTCOMES:
Maximum voluntary isometric contraction (MVIC) | Every time before the initiation of game(test time:1 seconds for each digit)
  Maximum voluntary isometric contraction (MVIC)

CONTACTS AND LOCATIONS:
Overall Officials: Fong-Chin Su, PHD, Principal Investigator — Chair Professor
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

REFERENCES:
- [Background] Bajaj S, Butler AJ, Drake D, Dhamala M. Brain effective connectivity during motor-imagery and execution following stroke and rehabilitation. Neuroimage Clin. 2015 Jun 28;8:572-82. doi: 10.1016/j.nicl.2015.06.006. eCollection 2015. PMID 26236627
- [Background] Polli A, Moseley GL, Gioia E, Beames T, Baba A, Agostini M, Tonin P, Turolla A. Graded motor imagery for patients with stroke: a non-randomized controlled trial of a new approach. Eur J Phys Rehabil Med. 2017 Feb;53(1):14-23. doi: 10.23736/S1973-9087.16.04215-5. Epub 2016 Jul 21. PMID 27442717
- [Background] Hsu HY, Chen PT, Kuan TS, Yang HC, Shieh SJ, Kuo LC. A Touch-Observation and Task-Based Mirror Therapy Protocol to Improve Sensorimotor Control and Functional Capability of Hands for Patients With Peripheral Nerve Injury. Am J Occup Ther. 2019 Mar/Apr;73(2):7302205020p1-7302205020p10. doi: 10.5014/ajot.2018.027763. PMID 30915963
- [Background] Ehrensberger M, Simpson D, Broderick P, Blake C, Horgan F, Hickey P, O'Reilly J, Monaghan K. Unilateral Strength Training and Mirror Therapy in Patients With Chronic Stroke: A Pilot Randomized Trial. Am J Phys Med Rehabil. 2019 Aug;98(8):657-665. doi: 10.1097/PHM.0000000000001162. PMID 31318745
- [Background] Dodakian L, Campbell Stewart J, Cramer SC. Motor imagery during movement activates the brain more than movement alone after stroke: a pilot study. J Rehabil Med. 2014 Oct;46(9):843-8. doi: 10.2340/16501977-1844. PMID 25182189
- [Background] Rossiter HE, Borrelli MR, Borchert RJ, Bradbury D, Ward NS. Cortical mechanisms of mirror therapy after stroke. Neurorehabil Neural Repair. 2015 Jun;29(5):444-52. doi: 10.1177/1545968314554622. Epub 2014 Oct 17. PMID 25326511
- [Background] Bello UM, Chan CCH, Winser SJ. Task Complexity and Image Clarity Facilitate Motor and Visuo-Motor Activities in Mirror Therapy in Post-stroke Patients. Front Neurol. 2021 Sep 22;12:722846. doi: 10.3389/fneur.2021.722846. eCollection 2021. PMID 34630297
- [Background] Ventoulis I, Gkouma KR, Ventouli S, Polyzogopoulou E. The Role of Mirror Therapy in the Rehabilitation of the Upper Limb's Motor Deficits After Stroke: Narrative Review. J Clin Med. 2024 Dec 20;13(24):7808. doi: 10.3390/jcm13247808. PMID 39768730
- [Background] Arya KN. Underlying neural mechanisms of mirror therapy: Implications for motor rehabilitation in stroke. Neurol India. 2016 Jan-Feb;64(1):38-44. doi: 10.4103/0028-3886.173622. PMID 26754990
- [Background] Formica C, De Salvo S, Muscara N, Bonanno L, Arcadi FA, Lo Buono V, Acri G, Quartarone A, Marino S. Applications of Near Infrared Spectroscopy and Mirror Therapy for Upper Limb Rehabilitation in Post-Stroke Patients: A Brain Plasticity Pilot Study. J Clin Med. 2024 Nov 4;13(21):6612. doi: 10.3390/jcm13216612. PMID 39518751
- [Background] Hamzei F, Lappchen CH, Glauche V, Mader I, Rijntjes M, Weiller C. Functional plasticity induced by mirror training: the mirror as the element connecting both hands to one hemisphere. Neurorehabil Neural Repair. 2012 Jun;26(5):484-96. doi: 10.1177/1545968311427917. Epub 2012 Jan 13. PMID 22247501
- [Background] Jaafar N, Che Daud AZ, Ahmad Roslan NF, Mansor W. Mirror Therapy Rehabilitation in Stroke: A Scoping Review of Upper Limb Recovery and Brain Activities. Rehabil Res Pract. 2021 Dec 31;2021:9487319. doi: 10.1155/2021/9487319. eCollection 2021. PMID 35003808
- [Background] Bello UM, Winser SJ, Chan CCH. Role of kinaesthetic motor imagery in mirror-induced visual illusion as intervention in post-stroke rehabilitation. Rev Neurosci. 2020 Aug 27;31(6):659-674. doi: 10.1515/revneuro-2019-0106. PMID 32229682
- [Background] Low E, Crewther SG, Ong B, Perre D, Wijeratne T. Compromised Motor Dexterity Confounds Processing Speed Task Outcomes in Stroke Patients. Front Neurol. 2017 Sep 21;8:484. doi: 10.3389/fneur.2017.00484. eCollection 2017. PMID 28983276
- [Background] Ao D, Song R, Tong KY. Sensorimotor control of tracking movements at various speeds for stroke patients as well as age-matched and young healthy subjects. PLoS One. 2015 Jun 1;10(6):e0128328. doi: 10.1371/journal.pone.0128328. eCollection 2015. PMID 26030289
- [Background] Gowda AS, Memon AN, Bidika E, Salib M, Rallabhandi B, Fayyaz H. Investigating the Viability of Motor Imagery as a Physical Rehabilitation Treatment for Patients With Stroke-Induced Motor Cortical Damage. Cureus. 2021 Mar 19;13(3):e14001. doi: 10.7759/cureus.14001. PMID 33884242
- [Background] Zich C, Ward NS, Forss N, Bestmann S, Quinn AJ, Karhunen E, Laaksonen K. Post-stroke changes in brain structure and function can both influence acute upper limb function and subsequent recovery. Neuroimage Clin. 2025;45:103754. doi: 10.1016/j.nicl.2025.103754. Epub 2025 Feb 13. PMID 39978147
- [Background] Lang CE, Schieber MH. Reduced muscle selectivity during individuated finger movements in humans after damage to the motor cortex or corticospinal tract. J Neurophysiol. 2004 Apr;91(4):1722-33. doi: 10.1152/jn.00805.2003. Epub 2003 Dec 10. PMID 14668295
- [Background] Ji EK, Wang HH, Jung SJ, Lee KB, Kim JS, Jo L, Hong BY, Lim SH. Graded motor imagery training as a home exercise program for upper limb motor function in patients with chronic stroke: A randomized controlled trial. Medicine (Baltimore). 2021 Jan 22;100(3):e24351. doi: 10.1097/MD.0000000000024351. PMID 33546067
- [Background] Lee SA, Cha HG. The effect of motor imagery and mirror therapy on upper extremity function according to the level of cognition in stroke patients. Int J Rehabil Res. 2019 Dec;42(4):330-336. doi: 10.1097/MRR.0000000000000366. PMID 31425348
- [Background] Li F, Zhang T, Li BJ, Zhang W, Zhao J, Song LP. Motor imagery training induces changes in brain neural networks in stroke patients. Neural Regen Res. 2018 Oct;13(10):1771-1781. doi: 10.4103/1673-5374.238616. PMID 30136692
- [Background] Hsu HY, Kuo LC, Lin YC, Su FC, Yang TH, Lin CW. Effects of a Virtual Reality-Based Mirror Therapy Program on Improving Sensorimotor Function of Hands in Chronic Stroke Patients: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2022 Jun;36(6):335-345. doi: 10.1177/15459683221081430. Epub 2022 Mar 28. PMID 35341360
- [Background] Park JY, Chang M, Kim KM, Kim HJ. The effect of mirror therapy on upper-extremity function and activities of daily living in stroke patients. J Phys Ther Sci. 2015 Jun;27(6):1681-3. doi: 10.1589/jpts.27.1681. Epub 2015 Jun 30. PMID 26180297
- [Background] Yavuzer G, Selles R, Sezer N, Sutbeyaz S, Bussmann JB, Koseoglu F, Atay MB, Stam HJ. Mirror therapy improves hand function in subacute stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2008 Mar;89(3):393-8. doi: 10.1016/j.apmr.2007.08.162. PMID 18295613
- [Background] Chan WC, Au-Yeung SSY. Recovery in the Severely Impaired Arm Post-Stroke After Mirror Therapy: A Randomized Controlled Study. Am J Phys Med Rehabil. 2018 Aug;97(8):572-577. doi: 10.1097/PHM.0000000000000919. PMID 29521681
- [Background] Wen X, Li L, Li X, Zha H, Liu Z, Peng Y, Liu X, Liu H, Yang Q, Wang J. Therapeutic Role of Additional Mirror Therapy on the Recovery of Upper Extremity Motor Function after Stroke: A Single-Blind, Randomized Controlled Trial. Neural Plast. 2022 Dec 31;2022:8966920. doi: 10.1155/2022/8966920. eCollection 2022. PMID 36624743
- [Background] Borges LR, Fernandes AB, Melo LP, Guerra RO, Campos TF. Action observation for upper limb rehabilitation after stroke. Cochrane Database Syst Rev. 2018 Oct 31;10(10):CD011887. doi: 10.1002/14651858.CD011887.pub2. PMID 30380586
- [Background] Fernandez-Solana J, Alvarez-Pardo S, Moreno-Villanueva A, Santamaria-Pelaez M, Gonzalez-Bernal JJ, Velez-Santamaria R, Gonzalez-Santos J. Efficacy of a Rehabilitation Program Using Mirror Therapy and Cognitive Therapeutic Exercise on Upper Limb Functionality in Patients with Acute Stroke. Healthcare (Basel). 2024 Feb 29;12(5):569. doi: 10.3390/healthcare12050569. PMID 38470680
- [Background] Corbetta D, Sarasso E, Agosta F, Filippi M, Gatti R. Mirror therapy for an adult with central post-stroke pain: a case report. Arch Physiother. 2018 Feb 23;8:4. doi: 10.1186/s40945-018-0047-y. eCollection 2018. PMID 29492272
- [Background] Iwanami J, Mutai H, Sagari A, Sato M, Kobayashi M. Relationship between Corticospinal Excitability While Gazing at the Mirror and Motor Imagery Ability. Brain Sci. 2023 Mar 9;13(3):463. doi: 10.3390/brainsci13030463. PMID 36979273
- [Background] Cengiz B, Vuralli D, Zinnuroglu M, Bayer G, Golmohammadzadeh H, Gunendi Z, Turgut AE, Irfanoglu B, Arikan KB. Analysis of mirror neuron system activation during action observation alone and action observation with motor imagery tasks. Exp Brain Res. 2018 Feb;236(2):497-503. doi: 10.1007/s00221-017-5147-5. Epub 2017 Dec 11. PMID 29230518
- [Background] Kang YJ, Ku J, Kim HJ, Park HK. Facilitation of corticospinal excitability according to motor imagery and mirror therapy in healthy subjects and stroke patients. Ann Rehabil Med. 2011 Dec;35(6):747-58. doi: 10.5535/arm.2011.35.6.747. Epub 2011 Dec 30. PMID 22506202
- [Background] Zhang K, Ding L, Wang X, Zhuang J, Tong S, Jia J, Guo X. Mirror therapy reduces excessive variability of motor network in stroke patients: a randomized controlled trial. Eur J Phys Rehabil Med. 2025 Apr;61(2):184-194. doi: 10.23736/S1973-9087.25.08844-6. Epub 2025 Apr 17. PMID 40243190
- [Background] Zhang H, Long Z, Ge R, Xu L, Jin Z, Yao L, Liu Y. Motor imagery learning modulates functional connectivity of multiple brain systems in resting state. PLoS One. 2014 Jan 17;9(1):e85489. doi: 10.1371/journal.pone.0085489. eCollection 2014. PMID 24465577
- [Background] Liu W, Cheng X, Rao J, Yu J, Lin Z, Wang Y, Wang L, Li D, Liu L, Gao R. Motor imagery therapy improved upper limb motor function in stroke patients with hemiplegia by increasing functional connectivity of sensorimotor and cognitive networks. Front Hum Neurosci. 2024 Feb 19;18:1295859. doi: 10.3389/fnhum.2024.1295859. eCollection 2024. PMID 38439937
- [Background] Thieme H, Morkisch N, Mehrholz J, Pohl M, Behrens J, Borgetto B, Dohle C. Mirror therapy for improving motor function after stroke. Cochrane Database Syst Rev. 2018 Jul 11;7(7):CD008449. doi: 10.1002/14651858.CD008449.pub3. PMID 29993119
- [Background] Abdullahi A, Wong TWL, Ng SSM. Rehabilitation of Severe Impairment in Motor Function after Stroke: Suggestions for Harnessing the Potentials of Mirror Neurons and the Mentalizing Systems to Stimulate Recovery. Brain Sci. 2022 Sep 28;12(10):1311. doi: 10.3390/brainsci12101311. PMID 36291245
- [Background] Garrison KA, Winstein CJ, Aziz-Zadeh L. The mirror neuron system: a neural substrate for methods in stroke rehabilitation. Neurorehabil Neural Repair. 2010 Jun;24(5):404-12. doi: 10.1177/1545968309354536. Epub 2010 Mar 5. PMID 20207851
- [Background] Wang J, Fritzsch C, Bernarding J, Krause T, Mauritz KH, Brunetti M, Dohle C. Cerebral activation evoked by the mirror illusion of the hand in stroke patients compared to normal subjects. NeuroRehabilitation. 2013;33(4):593-603. doi: 10.3233/NRE-130999. PMID 24018372
- [Background] Zhang K, Ding L, Wang X, Zhuang J, Tong S, Jia J, Guo X. Evidence of mirror therapy for recruitment of ipsilateral motor pathways in stroke recovery: A resting fMRI study. Neurotherapeutics. 2024 Mar;21(2):e00320. doi: 10.1016/j.neurot.2024.e00320. Epub 2024 Jan 22. PMID 38262102
- [Background] Bai Z, Zhang J, Zhang Z, Shu T, Niu W. Comparison Between Movement-Based and Task-Based Mirror Therapies on Improving Upper Limb Functions in Patients With Stroke: A Pilot Randomized Controlled Trial. Front Neurol. 2019 Mar 26;10:288. doi: 10.3389/fneur.2019.00288. eCollection 2019. PMID 30972016
- [Background] Schaefer SY, DeJong SL, Cherry KM, Lang CE. Grip type and task goal modify reach-to-grasp performance in post-stroke hemiparesis. Motor Control. 2012 Apr;16(2):245-64. doi: 10.1123/mcj.16.2.245. Epub 2012 Feb 16. PMID 22357103
- [Background] Kang N, Cauraugh JH. Force control in chronic stroke. Neurosci Biobehav Rev. 2015 May;52:38-48. doi: 10.1016/j.neubiorev.2015.02.005. Epub 2015 Feb 19. PMID 25704075
- [Background] Wriessnegger SC, Kirchmeyr D, Bauernfeind G, Muller-Putz GR. Force related hemodynamic responses during execution and imagery of a hand grip task: A functional near infrared spectroscopy study. Brain Cogn. 2017 Oct;117:108-116. doi: 10.1016/j.bandc.2017.06.010. Epub 2017 Jun 30. PMID 28673464
- [Background] Spraker MB, Corcos DM, Vaillancourt DE. Cortical and subcortical mechanisms for precisely controlled force generation and force relaxation. Cereb Cortex. 2009 Nov;19(11):2640-50. doi: 10.1093/cercor/bhp015. Epub 2009 Mar 2. PMID 19254959
- [Background] Paclet F, Quaine F. Motor control theories improve biomechanical model of the hand for finger pressing tasks. J Biomech. 2012 Apr 30;45(7):1246-51. doi: 10.1016/j.jbiomech.2012.01.038. Epub 2012 Feb 20. PMID 22356843
- [Background] Aderinto N, AbdulBasit MO, Olatunji G, Adejumo T. Exploring the transformative influence of neuroplasticity on stroke rehabilitation: a narrative review of current evidence. Ann Med Surg (Lond). 2023 Aug 7;85(9):4425-4432. doi: 10.1097/MS9.0000000000001137. eCollection 2023 Sep. PMID 37663728
- [Background] Takeuchi N, Izumi S. Rehabilitation with poststroke motor recovery: a review with a focus on neural plasticity. Stroke Res Treat. 2013;2013:128641. doi: 10.1155/2013/128641. Epub 2013 Apr 30. PMID 23738231
- [Background] Amin F, Waris A, Syed S, Amjad I, Umar M, Iqbal J, Omer Gilani S. Effectiveness of Immersive Virtual Reality-Based Hand Rehabilitation Games for Improving Hand Motor Functions in Subacute Stroke Patients. IEEE Trans Neural Syst Rehabil Eng. 2024;32:2060-2069. doi: 10.1109/TNSRE.2024.3405852. Epub 2024 May 30. PMID 38801680
- [Background] Gnanaprakasam A, Karthikbabu S, Ravishankar N, Solomon JM. Effect of task-based bilateral arm training on upper limb recovery after stroke: A systematic review and meta-analysis. J Stroke Cerebrovasc Dis. 2023 Jul;32(7):107131. doi: 10.1016/j.jstrokecerebrovasdis.2023.107131. Epub 2023 May 4. PMID 37148628
- [Background] Akter R, Sharma N, Ahmed S, Srivastav AK. Combined effect of Brunnstrom's hand rehabilitation and functional electrical stimulation for improving hand function in patients with chronic stroke: A randomized controlled trial. J Bodyw Mov Ther. 2023 Jul;35:84-90. doi: 10.1016/j.jbmt.2023.04.021. Epub 2023 Apr 28. PMID 37330808
- [Background] Lee HC, Kuo FL, Lin YN, Liou TH, Lin JC, Huang SW. Effects of Robot-Assisted Rehabilitation on Hand Function of People With Stroke: A Randomized, Crossover-Controlled, Assessor-Blinded Study. Am J Occup Ther. 2021 Jan-Feb;75(1):7501205020p1-7501205020p11. doi: 10.5014/ajot.2021.038232. PMID 33399050
- [Background] Smedes F, Giacometti da Silva L. Motor learning with the PNF-concept, an alternative to constrained induced movement therapy in a patient after a stroke; a case report. J Bodyw Mov Ther. 2019 Jul;23(3):622-627. doi: 10.1016/j.jbmt.2018.05.003. Epub 2018 May 31. PMID 31563380
- [Background] Maggio MG, Latella D, Maresca G, Sciarrone F, Manuli A, Naro A, De Luca R, Calabro RS. Virtual Reality and Cognitive Rehabilitation in People With Stroke: An Overview. J Neurosci Nurs. 2019 Apr;51(2):101-105. doi: 10.1097/JNN.0000000000000423. PMID 30649091
- [Background] Aisen ML, Krebs HI, Hogan N, McDowell F, Volpe BT. The effect of robot-assisted therapy and rehabilitative training on motor recovery following stroke. Arch Neurol. 1997 Apr;54(4):443-6. doi: 10.1001/archneur.1997.00550160075019. PMID 9109746
- [Background] Kim BR, Chun MH, Kim LS, Park JY. Effect of virtual reality on cognition in stroke patients. Ann Rehabil Med. 2011 Aug;35(4):450-9. doi: 10.5535/arm.2011.35.4.450. Epub 2011 Aug 31. PMID 22506159
- [Background] Taub E, Wolf SL. Constraint Induced Movement Techniques To Facilitate Upper Extremity Use in Stroke Patients. Top Stroke Rehabil. 1997 Jan;3(4):38-61. doi: 10.1080/10749357.1997.11754128. PMID 27620374
- [Background] Altschuler EL, Wisdom SB, Stone L, Foster C, Galasko D, Llewellyn DM, Ramachandran VS. Rehabilitation of hemiparesis after stroke with a mirror. Lancet. 1999 Jun 12;353(9169):2035-6. doi: 10.1016/s0140-6736(99)00920-4. No abstract available. PMID 10376620
- [Background] Liew SL, Schweighofer N, Cole JH, Zavaliangos-Petropulu A, Tavenner BP, Han LKM, Hahn T, Schmaal L, Donnelly MR, Jeong JN, Wang Z, Abdullah A, Kim JH, Hutton A, Barisano G, Borich MR, Boyd LA, Brodtmann A, Buetefisch CM, Byblow WD, Cassidy JM, Charalambous CC, Ciullo V, Conforto AB, Dacosta-Aguayo R, DiCarlo JA, Domin M, Dula AN, Egorova-Brumley N, Feng W, Geranmayeh F, Gregory CM, Hanlon CA, Hayward K, Holguin JA, Hordacre B, Jahanshad N, Kautz SA, Khlif MS, Kim H, Kuceyeski A, Lin DJ, Liu J, Lotze M, MacIntosh BJ, Margetis JL, Mataro M, Mohamed FB, Olafson ER, Park G, Piras F, Revill KP, Roberts P, Robertson AD, Sanossian N, Schambra HM, Seo NJ, Soekadar SR, Spalletta G, Stinear CM, Taga M, Tang WK, Thielman GT, Vecchio D, Ward NS, Westlye LT, Winstein CJ, Wittenberg GF, Wolf SL, Wong KA, Yu C, Cramer SC, Thompson PM. Association of Brain Age, Lesion Volume, and Functional Outcome in Patients With Stroke. Neurology. 2023 May 16;100(20):e2103-e2113. doi: 10.1212/WNL.0000000000207219. Epub 2023 Apr 4. PMID 37015818
- [Background] Mawase F, Cherry-Allen K, Xu J, Anaya M, Uehara S, Celnik P. Pushing the Rehabilitation Boundaries: Hand Motor Impairment Can Be Reduced in Chronic Stroke. Neurorehabil Neural Repair. 2020 Aug;34(8):733-745. doi: 10.1177/1545968320939563. PMID 32845230
- [Background] Lodha N, Naik SK, Coombes SA, Cauraugh JH. Force control and degree of motor impairments in chronic stroke. Clin Neurophysiol. 2010 Nov;121(11):1952-61. doi: 10.1016/j.clinph.2010.04.005. PMID 20435515
- [Background] Yamawaki N, Raineri Tapies MG, Stults A, Smith GA, Shepherd GM. Circuit organization of the excitatory sensorimotor loop through hand/forelimb S1 and M1. Elife. 2021 Apr 14;10:e66836. doi: 10.7554/eLife.66836. PMID 33851917
- [Background] Codol O, Kashefi M, Forgaard CJ, Galea JM, Pruszynski JA, Gribble PL. Sensorimotor feedback loops are selectively sensitive to reward. Elife. 2023 Jan 13;12:e81325. doi: 10.7554/eLife.81325. PMID 36637162
- [Background] Bolognini N, Russo C, Edwards DJ. The sensory side of post-stroke motor rehabilitation. Restor Neurol Neurosci. 2016 Apr 11;34(4):571-86. doi: 10.3233/RNN-150606. PMID 27080070
- [Background] Meyer S, Karttunen AH, Thijs V, Feys H, Verheyden G. How do somatosensory deficits in the arm and hand relate to upper limb impairment, activity, and participation problems after stroke? A systematic review. Phys Ther. 2014 Sep;94(9):1220-31. doi: 10.2522/ptj.20130271. Epub 2014 Apr 24. PMID 24764072
- [Background] Raghavan P, Santello M, Gordon AM, Krakauer JW. Compensatory motor control after stroke: an alternative joint strategy for object-dependent shaping of hand posture. J Neurophysiol. 2010 Jun;103(6):3034-43. doi: 10.1152/jn.00936.2009. Epub 2010 Mar 24. PMID 20457866
- [Background] Eschmann H, Heroux ME, Cheetham JH, Potts S, Diong J. Thumb and finger movement is reduced after stroke: An observational study. PLoS One. 2019 Jun 12;14(6):e0217969. doi: 10.1371/journal.pone.0217969. eCollection 2019. PMID 31188859
- [Background] Ruan Y, Shin H, Hu X. Quantifying Muscle Co-Activation for Impaired Finger Independence in Stroke Survivors. IEEE Trans Biomed Eng. 2024 Nov;71(11):3293-3301. doi: 10.1109/TBME.2024.3416908. Epub 2024 Oct 25. PMID 38896507
- [Background] Lang CE, DeJong SL, Beebe JA. Recovery of thumb and finger extension and its relation to grasp performance after stroke. J Neurophysiol. 2009 Jul;102(1):451-9. doi: 10.1152/jn.91310.2008. Epub 2009 May 20. PMID 19458140
- [Background] O'Dwyer NJ, Ada L, Neilson PD. Spasticity and muscle contracture following stroke. Brain. 1996 Oct;119 ( Pt 5):1737-49. doi: 10.1093/brain/119.5.1737. PMID 8931594
- [Background] Lee SW, Qiu D, Fischer HC, Conrad MO, Kamper DG. Modulation of finger muscle activation patterns across postures is coordinated across all muscle groups. J Neurophysiol. 2020 Aug 1;124(2):330-341. doi: 10.1152/jn.00088.2020. Epub 2020 Jun 24. PMID 32579416
- [Background] Jorgensen HS, Nakayama H, Raaschou HO, Vive-Larsen J, Stoier M, Olsen TS. Outcome and time course of recovery in stroke. Part II: Time course of recovery. The Copenhagen Stroke Study. Arch Phys Med Rehabil. 1995 May;76(5):406-12. doi: 10.1016/s0003-9993(95)80568-0. PMID 7741609
- [Background] Sahrizan NSA, Yahya N, Law ZK, Wan Zaidi WA, Nabilah Ismail U, Afifah NH, Azri A, Abdul Manan H. A systematic review of alterations in sensorimotor networks following stroke: implications for integration and functional outcomes across recovery stages. Front Neurol. 2025 May 27;16:1456146. doi: 10.3389/fneur.2025.1456146. eCollection 2025. PMID 40496121
- [Background] Buetefisch CM, Revill KP, Haut MW, Kowalski GM, Wischnewski M, Pifer M, Belagaje SR, Nahab F, Cobia DJ, Hu X, Drake D, Hobbs G. Abnormally reduced primary motor cortex output is related to impaired hand function in chronic stroke. J Neurophysiol. 2018 Oct 1;120(4):1680-1694. doi: 10.1152/jn.00715.2017. Epub 2018 Jun 20. PMID 29924707
- [Background] Lai SM, Studenski S, Duncan PW, Perera S. Persisting consequences of stroke measured by the Stroke Impact Scale. Stroke. 2002 Jul;33(7):1840-4. doi: 10.1161/01.str.0000019289.15440.f2. PMID 12105363
- [Background] Gilbert CD, Sigman M. Brain states: top-down influences in sensory processing. Neuron. 2007 Jun 7;54(5):677-96. doi: 10.1016/j.neuron.2007.05.019. PMID 17553419
- [Background] Ward NS, Newton JM, Swayne OB, Lee L, Frackowiak RS, Thompson AJ, Greenwood RJ, Rothwell JC. The relationship between brain activity and peak grip force is modulated by corticospinal system integrity after subcortical stroke. Eur J Neurosci. 2007 Mar;25(6):1865-73. doi: 10.1111/j.1460-9568.2007.05434.x. PMID 17432972
- [Background] Kim HW, Lee DG. Resting-State Metabolism of Hand Knob Area on 18F-FDG PET-CT According to Hand Function and Tractography of Corticospinal Tract After Stroke. Ann Rehabil Med. 2017 Apr;41(2):171-177. doi: 10.5535/arm.2017.41.2.171. Epub 2017 Apr 27. PMID 28503448
- [Background] Edin BB, Westling G, Johansson RS. Independent control of human finger-tip forces at individual digits during precision lifting. J Physiol. 1992 May;450:547-64. doi: 10.1113/jphysiol.1992.sp019142. PMID 1432717
- [Background] Ambike SS, Paclet F, Latash ML, Zatsiorsky VM. Grip-force modulation in multi-finger prehension during wrist flexion and extension. Exp Brain Res. 2013 Jun;227(4):509-22. doi: 10.1007/s00221-013-3527-z. Epub 2013 Apr 30. PMID 23625077
- [Background] Li L, Scott CA, Rothwell PM. Association of Younger vs Older Ages With Changes in Incidence of Stroke and Other Vascular Events, 2002-2018. JAMA. 2022 Aug 9;328(6):563-574. doi: 10.1001/jama.2022.12759. PMID 35943470
- [Background] Pu L, Wang L, Zhang R, Zhao T, Jiang Y, Han L. Projected Global Trends in Ischemic Stroke Incidence, Deaths and Disability-Adjusted Life Years From 2020 to 2030. Stroke. 2023 May;54(5):1330-1339. doi: 10.1161/STROKEAHA.122.040073. Epub 2023 Apr 24. PMID 37094034
- [Background] Hsieh FI, Chiou HY. Stroke: morbidity, risk factors, and care in taiwan. J Stroke. 2014 May;16(2):59-64. doi: 10.5853/jos.2014.16.2.59. Epub 2014 May 30. PMID 24949310
- [Background] Unnithan AKA, Das JM. Hemorrhagic Stroke. 2025 Dec 13. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK559173/ PMID 32644599
- [Background] Lui F, Khan Suheb MZ, Patti L. Ischemic Stroke. 2025 Feb 21. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK499997/ PMID 29763173
- [Background] Cheng Y, Lin Y, Shi H, Cheng M, Zhang B, Liu X, Shi C, Wang Y, Xia C, Xie W. Projections of the Stroke Burden at the Global, Regional, and National Levels up to 2050 Based on the Global Burden of Disease Study 2021. J Am Heart Assoc. 2024 Dec 3;13(23):e036142. doi: 10.1161/JAHA.124.036142. Epub 2024 Nov 22. PMID 39575720
- [Background] Inchai P, Tsai WC, Chiu LT, Kung PT. Incidence, risk, and associated risk factors of stroke among people with different disability types and severities: A national population-based cohort study in Taiwan. Disabil Health J. 2021 Oct;14(4):101165. doi: 10.1016/j.dhjo.2021.101165. Epub 2021 Jul 3. PMID 34266788
- [Background] Zhu L, Fratiglioni L, Guo Z, Aguero-Torres H, Winblad B, Viitanen M. Association of stroke with dementia, cognitive impairment, and functional disability in the very old: a population-based study. Stroke. 1998 Oct;29(10):2094-9. doi: 10.1161/01.str.29.10.2094. PMID 9756588
- [Background] GBD 2021 Stroke Risk Factor Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2021: a systematic analysis for the Global Burden of Disease Study 2021. Lancet Neurol. 2024 Oct;23(10):973-1003. doi: 10.1016/S1474-4422(24)00369-7. PMID 39304265